CLINICAL TRIAL: NCT00749450
Title: Short Course Oncology Therapy - A Study of Adjuvant Chemotherapy in Colorectal Cancer
Brief Title: Combination Chemotherapy After Surgery in Treating Patients With High-Risk Stage II or Stage III Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Research UK, Glasgow (Other)
Responsible Party: Principal Investigator, Laura Alexander, Project Manager, Cancer Research UK, Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000613042; CRUK-SCOT; ISRCTN59757862; EudraCT 2007-003957-10; EU-20874; SCOT-2007-01
Record Dates: First submitted 2008-09-06; First posted 2008-09-09 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive OxMdG or XELOX combination chemotherapy for a total of 12 courses for treatment lasting a total of 24 weeks.
  Interventions: Drug: capecitabine; Drug: fluorouracil; Drug: oxaliplatin
- Arm II (Experimental): Patients receive OxMdG or XELOX combination chemotherapy for a total of 6 courses for treatment lasting a total of 12 weeks.
  Interventions: Drug: capecitabine; Drug: fluorouracil; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine — Given orally
Drug: fluorouracil — Given IV
Drug: oxaliplatin — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, fluorouracil, and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known which combination chemotherapy regimen is more effective in treating patients who have undergone surgery for high-risk colorectal cancer.

PURPOSE: This randomized phase III trial is studying chemotherapy given after surgery in treating patients with high-risk stage II or stage III colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the efficacy and compare the associated toxicity of adjuvant chemotherapy lasting 12 weeks vs 24 weeks in patients with fully resected high-risk stage II or III colorectal cancer.
* To conduct an economic analysis of the cost effectiveness of these regimens.
* To compare the randomization methodologies used in this study.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center's recruitment potential. Patients are randomized (within 10 weeks after surgery and before or after receiving 12 weeks of chemotherapy) to 1 of 2 treatment arms. The treatment regimen that a patient receives (Oxaliplatin Modified DeGramont [OxMdG] or XELOX) is determined by the participating center.

* Arm I: Patients receive 12 courses of OxMdG (described below) or XELOX (described below)combination chemotherapy (6 additional courses if patient already received 6 courses) for treatment lasting a total of 24 weeks.
* Arm II: Patients receive 6 courses of OxMdG or XELOX combination chemotherapy (no additional courses if patient already received 6 courses) for treatment lasting a total of 12 weeks.

The two adjuvant combination chemotherapy regimens are administered as follows:

* OxMdG: Patients receive oxaliplatin IV over 2 hours and fluorouracil IV continuously over 46 hours on day 1. Treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* XELOX: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of-life assessments periodically using the EORTC QLQ-C30, EORTC QLQ-CR29, EQ-5D, and GOG Ntx4 questionnaires.

After completion of study treatment, patients are followed periodically for up to 7 years.

Peer Reviewed and Funded by Medical Research Council (MRC)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal cancer meeting 1 of the following criteria:

  * High-risk stage IIB disease, defined as T4 disease, perforation, obstruction, < 10 nodes examined, poorly differentiated histology, extramural venous invasion, or extramural lymphatic invasion
  * Fully resected stage III disease
* Patients with rectal cancer must meet the following criteria:

  * Underwent prior total mesorectal excision surgery with negative resection (R0) margins
  * No prior pre-operative or scheduled post-operative combined chemotherapy and radiotherapy
* No evidence of residual or metastatic disease
* Deemed suitable for adjuvant chemotherapy

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy > 5 years with reference to noncancer-related diseases
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Carcinoembryonic antigen (CEA) levels normal
* Glomerular filtration rate ≥ 30 mL/min (no moderate or severe renal impairment)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must effective contraception
* More than 12 months since prior and no active clinically significant cardiovascular disease, including any of the following:

  * Cerebrovascular accident
  * Myocardial infarction
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Uncontrolled hypertension (i.e., blood pressure > 150/100 mm Hg)
* Disease-free interval of ≥ 5 years for previous malignancy other than adequately treated in situ carcinoma of the uterine cervix or basal cell or squamous cell carcinoma of the skin
* No known or suspected dihydropyrimidine dehydrogenase deficiency

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No more than 10 weeks since prior surgery and recovered
* No prior chemotherapy (except in patients randomized after 12 weeks of adjuvant therapy)
* No prior abdomino-pelvic radiotherapy, with the exception of short-course pre-operative radiotherapy for rectal cancer
* No concurrent brivudine or sorivudine for patients taking capecitabine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6088 (Actual)
Dates: Start 2008-03; Primary Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years

SECONDARY OUTCOMES:
Overall survival | assessed during 5 year recruitment period and maximum 7 year follow up period
Cost-effectiveness | assessed during 5 year recruitment period
Toxicity according to NCI CTCAE Version 3.0 | assessed during 5 year recruitment period
Quality of life as assessed by EORTC QLQ-C30, EORTC QLQ-CR29, EQ-5D, and GOG Ntx4 | assessed during 5 year recruitment period

CONTACTS AND LOCATIONS:
Overall Officials: Tim Iveson, FRCP, MD, MRCP, MBBS, BSC, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Gallois C, Shi Q, Meyers JP, Iveson T, Alberts SR, de Gramont A, Sobrero AF, Haller DG, Oki E, Shields AF, Goldberg RM, Kerr R, Lonardi S, Yothers G, Kelly C, Boukovinas I, Labianca R, Sinicrope FA, Souglakos I, Yoshino T, Meyerhardt JA, Andre T, Papamichael D, Taieb J. Prognostic Impact of Early Treatment and Oxaliplatin Discontinuation in Patients With Stage III Colon Cancer: An ACCENT/IDEA Pooled Analysis of 11 Adjuvant Trials. J Clin Oncol. 2023 Feb 1;41(4):803-815. doi: 10.1200/JCO.21.02726. Epub 2022 Oct 28. PMID 36306483
- [Derived] Iveson TJ, Sobrero AF, Yoshino T, Souglakos I, Ou FS, Meyers JP, Shi Q, Grothey A, Saunders MP, Labianca R, Yamanaka T, Boukovinas I, Hollander NH, Galli F, Yamazaki K, Georgoulias V, Kerr R, Oki E, Lonardi S, Harkin A, Rosati G, Paul J. Duration of Adjuvant Doublet Chemotherapy (3 or 6 months) in Patients With High-Risk Stage II Colorectal Cancer. J Clin Oncol. 2021 Feb 20;39(6):631-641. doi: 10.1200/JCO.20.01330. Epub 2021 Jan 13. PMID 33439695